CLINICAL TRIAL: NCT02838121
Title: Investigation on the Prevention of Periprosthetic Bone Loss After Total Hip Replacement by Annual Bisphosphonate Therapy: A Prospective Randomized Clinical Trial
Brief Title: Prevention of Periprosthetic Bone Loss After Total Hip Replacement by Annual Bisphosphonate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mel Shiuann-Sheng Lee (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Mel Shiuann-Sheng Lee, Clinical Professor, Chang Gung Memorial Hospital, Department of Orthopaedic Surgery, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98-1150A3
Record Dates: First submitted 2016-07-07; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Prevention of BMD Loss After THR; Serum Markers of Bone Turnover; Functional Outcomes
Keywords: bisphosphonate; Total hip replacement; functional outcomes; bone mineral density
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclasta (Experimental): Aclasta IV once annual for 2 years
  Interventions: Drug: Aclasta
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclasta — Aclasta once annually for 2 years
  Arms: Aclasta
Drug: Placebo — No IV aclasta
  Arms: Placebo

SUMMARY:
Periprosthetic bone loss caused by stress-shielding effect, a phenomenon of bone atrophy under mechanical unloading after THR implantation, further compromises the longevity of implant. The prospective randomized study is aimed to investigate the periprosthetic bone loss after primary total hip replacements.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open-label clinical trial. The study will be performed in patients after obtaining informed consent. Group assignment is by drawing a sealed envelops based on random table. (1) Group 1: Experimental group 30 cases, Aclasta® (Zoledronic acid 5mg/100ml) is given intravenously on the 4th postoperative day and one year after the total hip replacement, (2) Group 2: Control group, 30 cases, no bisphosphonate is given to the patients. Only the unilateral coxarthrosis will be recruited for the study. Patients will be analyzed with (1) DXA study (2) Clinical assessment (Harris hip score and SF-12) (3) X-ray (4) serum marker of bone turnover. Patients will be scheduled for specified examinations preoperatively, postoperatively 6 weeks, 3 months, 6 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female,between 35 and 85 years of age
2. Indicated for Total hip replacement for various hip diseases
3. Has preoperative DXA study within 3 months before the total hip replacement procedure or willing to receive preoperative DXA study as a baseline comparison
4. Signed written informed consent
5. Standard transgluteal approach for total hip replacement using Zimmer Triology Cup and Versys Fiber Metal Taper Stem with metal to highly cross-linked polyethylene bearing surface

Exclusion Criteria:

1. Any prior use of intravenous bisphosphonate within the last 2 years
2. Uncontrolled seizure disorders associated with falls
3. A history of invasive malignancy of any organ system, treated or untreated, within the past five years; excluding, basal cell or squamous cell carcinoma of the skin, colonic polyps with non-invasive malignancy which have been removed
4. Carcinoma in situ of the uterine cervix
5. History of osteogenesis imperfecta, multiple myeloma, or Paget's disease
6. Active primary hyperparathyroidism
7. History of iritis or uveitis
8. Self-reported history of diabetic nephropathy or retinopathy
9. AST or ALT more than twice the upper limit of normal
10. Alkaline phosphatase more than twice the upper limit of normal
11. Serum calcium 2.75 mmol/L (11.0 mg/dL)
12. Baseline renal insufficiency (calculated creatinine clearance 35 ml/min)
13. History of hypersensitivity to bisphosphonates
14. Use of any investigational drug(s) and/or devices within 30 days prior to randomization
15. Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from adhering to the Protocol or completing the trial per protocol
16. Use of hip protectors
17. With implant or prosthesis on the contralateral hip joint

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
bone mineral density [g/cm2] of the 7 Gruen zones | 5 years
  bone mineral density measured by dual energy x-ray absorptiometry
bone mineral density change relative to the baseline values of the 7 Gruen zones | 5 years
  bone mineral density measured by dual energy x-ray absorptiometry
implant loosening or migration | 5 years
  check the implant position by serial standard X ray follow-up

SECONDARY OUTCOMES:
serum alkaline phosphatase | 5 years
serum calcium level | 5 years
serum phosphate level | 5 years
serum osteocalcin level | 5 years
serum N-telopeptide procollagen level | 5 years
serum creatinine level | 5 years
  renal function and glomerular filtration rate
serum alanine aminotransferase level | 5 years
  liver function
serum aspartate aminotransferase level | 5 years
  liver function
harris hip score | 5 years
  hip function measurement
short form-12 | 5 years
  life quality measurement
University of California Los Angeles Activity Score | 5 years
  functional and activity evaluation, 10 point scale

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kweishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Chang Gung Memorial Hospital — http://www.cgmh.org.tw
- See also: American Academy of Orthopaedic Surgeons — http://www.AAOS.org